CLINICAL TRIAL: NCT05830487
Title: Effect of Dietary Intervention on Serum Advanced Glycation End Products and Metabolic Profile in Polycystic Ovary Syndrome Patients
Brief Title: Advanced Glycation End Products and Dietary Intervention in Polycystic Ovary Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Merve Özdemir, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HACETTEPE UNIVERSITY-OZDEMIR-1
Record Dates: First submitted 2023-01-25; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Polycystic Ovary Syndrome; Diet Habit
Keywords: advanced glycation end products; diet
MeSH Terms: conditions — Polycystic Ovary Syndrome; Feeding Behavior | interventions — CD36 Antigens

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low AGE diet with reduced energy and fat (Experimental): Low advanced glycation end products diet with reduced energy and fat
  Interventions: Behavioral: Low AGE diet with reduced energy and fat
- Energy and fat-reduced normal diet (Experimental): only energy and fat-reduced diet, advanced glycation end products intake will not be interfered with.
  Interventions: Behavioral: Energy and fat-reduced normal diet

INTERVENTIONS:
Behavioral: Low AGE diet with reduced energy and fat — This group will be given a low AGE diet with reduced energy and fat,.
  Arms: Low AGE diet with reduced energy and fat
Behavioral: Energy and fat-reduced normal diet — This group will be given a diet with reduced energy and fat, and AGE levels will not be interfered with
  Arms: Energy and fat-reduced normal diet

SUMMARY:
Recently, the negative effects of advanced glycation end products on the pathophysiology of some diseases have attracted attention. This study was planned to evaluate the effect of dietary intervention and weight loss on serum advanced glycation and disease pathogenesis in patients with polycystic ovary syndrome.

DETAILED DESCRIPTION:
The significantly increased consumption of processed foods in recent years has also increased the amount of sugar and fat in the diet. These changes in dietary habits also increase exposure to advanced glycation end products. Advanced glycation end products (AGEs) are the products occurred as a result of the Maillard reaction by the combination of the carbonyl group of carbohydrates and the free amino groups of amino acids. Advance glycation end products causes irreversible cross-linking of proteins, resulting in loss of protein structure and function. Advanced glycation end products formation is a slow process in normal conditions, but chronic diseases such as diabetes, insulin resistance, aging, oxidative stress and PCOS accelerate the occurrence of endogenous AGEs.

Polycystic ovary syndrome (PCOS) is an endocrine disorder that is characterized by hyperandrogenism, oligo/anovulation and polycystic ovaries and it affects up to 25% of reproductive-aged women. Women with PCOS have been shown to have an increase in the levels of AGEs in the bloodstream and the expression of proinflammatory receptors of AGEs in the ovaries, such as RAGE. In addition, the levels of protective anti-inflammatory receptors called soluble receptors for advanced glycation end products (sRAGE) were found to be low in women with PCOS. Patient with PCOS in particular have high levels of serum AGEs, regardless of their body weight or the presence of insulin resistance.

In this project, aimed to investigate effect of a diet with reduced energy and fat content and a low AGE diet with reduced energy and fat content for 12 weeks in overweight and obese individuals with polycystic ovary syndrome.

Body composition, anthropometric measurements, serum AGE levels, serum antioxidant capacity, inflammation, cardio metabolic profile, hormonal profile, and also Anti-Mullerian Hormone (AMH) values will be examined in individuals and the results will be evaluated by comparing diet groups. Volunteers participating in the study will apply one of two different dietary treatments to be determined by stratified randomization method for 12 weeks. The smallest sample size was calculated as a total of 24 patients, 12 patients in each intervention group, taking into account the change in serum AGE value at 80% power and 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:• Being diagnosed with PCOS Being between the ages of 19-35 Having a body mass index of more than 25 kg/m2 Volunteering to work

-

Exclusion Criteria:

* Presence of chronic disease (Diabetes, Hypertension, Atherosclerotic heart diseases, gastrointestinal system diseases..)

  * Being in pregnancy-lactation or menopause period
  * Using oral contraceptive medication
  * Using vitamin-mineral support
  * Receiving a special dietary treatment
  * To have applied a weight loss diet in the last 3 months
  * To smoke

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Serum advanced glycation end products levels | 12 weeks
  The comparison of serum advanced glycation end products levels of 24 patients before and after dietary intervention
Total antioxidant/oxidant capacity | 12 weeks
  The comparison total antioxidant/oxidant capacity levels of 24 patients before and after dietary intervention
İnflammation | 12 weeks
  The comparison tnf-a and hs-CRP levels of 24 patients before and after dietary intervention
Cardio metabolic profile | 12 weeks
  The comparison of fasting insulin (mg/dL), fasting blood sugar (mg/dL), lipid parameters (triglyceride (mg/dL), LDL-C (mg/dL), HDL-C (mg/dL), total cholesterol (mg/dL)) values of 24 patients at baseline and week 12.
Hormonal Profile | 12 weeks
  From hormonal indicators total testosterone (ng/mL), sex hormone-binding globulin ng/mL) , Anti mullerian hormone (ng/mL) values of 24 patients at baseline and week 12 will be compared.

SECONDARY OUTCOMES:
Body composition | 12 weeks
  The comparison of body fat percentage of 24 patients at baseline and week 12
Body weight | 12 weeks
  The comparison of body weight (kg) of 24 patients at baseline and week 12
Body Mass İndex | 12 weeks
  Body mass index (kg/m^2) of 24 patients at baseline and week 12 will be compared
Circumference measurements | 12 weeks
  waist circumference (cm) and hip circumference (cm) of 24 patients at baseline and week 12 will be compared

CONTACTS AND LOCATIONS:
Overall Officials: merve özdemir, Principal Investigator — researcher
Locations (1):
- hacettepe University, Ankara, Altindag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozdemir M, Mumusoglu S, Bilgic P. Comparison of Metabolic and Hormonal Profiles between Low-Advanced Glycation End Products (AGEs) and Standard AGEs-Containing Weight-Loss Diets in Overweight Phenotype-A PCOS Patients: A Randomized Clinical Trial. Reprod Sci. 2025 Apr;32(4):1190-1201. doi: 10.1007/s43032-025-01808-8. Epub 2025 Feb 14. PMID 39953370